CLINICAL TRIAL: NCT03144011
Title: Early Diagnosis of Acute Kidney Injury in Children With Congenital Heart Disease After Cardiopulmonary Bypass
Brief Title: Acute Kidney Injury in Children After Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Other Study IDs: 20.03 №194
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Congenital Heart Disease in Children; Cardiopulmonary Bypass
Keywords: acute kidney injury, cardiosurgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is a common complication in patients with congenital heart defects after cardiopulmonary bypass. The death rate from AKI in critically ill children remains high and reaches 60%.

The basic criteria for diagnosing and assessing the severity of kidney injury until recently were the level of serum creatinine and the amount of urine released. However, it should be noted that the level of serum creatinine, traditionally used to assess renal function, does not significantly increase until a decrease of more than 50% of the glomerular filtration rate, in addition, its level depends also on some extrarenal causes. Artificial blood circulation and hemodilution leads to the preservation of the level of creatinine at sufficiently low levels up to 1-3 days postoperative period. The level of diuresis as well as the level of creatinine is a nonspecific criterion after cardiac surgery and depends on several factors.

Currently, in the field of acute renal injury studies, progress has been made in the emergence of new biomarkers such as the tissue inhibitor metalloproteinase-2 (TIMP-2) and insulin-like growth factor binding globulin-7 (IGFBP7), which are early markers of acute renal damage. In a study in adult patients, it was shown that the levels of TIMP-2 and IGFBP7 increased In the first 24-48 before the diagnosis of IR-associated renal damage.

Among pediatric patients with congenital heart defects, such studies are single and only present for the age group 3 and older, which also demonstrated the high specificity and prognostic significance of these biomarkers in the early diagnosis of acute renal damage.

It should also be noted that, in spite of the high specificity of the markers described, it is also necessary to note their considerable cost.

Thus, taking into account the above, it is planned to compare and identify the relationship of these indicators with such parameter as the index of renal vascular resistance, the increase of which in the pre- and postoperative period may serve as a sign of the beginning acute renal injury.

ELIGIBILITY:
Inclusion Criteria:

Age from 1 month to 1 year Presence of congenital heart disease Radical correction of the defect in conditions of cardiopulmonary bypass

Exclusion Criteria:

Inconsistency with age criteria Cardiotonic support before surgery Acute renal, acute liver failure before surgery

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 1 month to 1 year with congenital heart disease, operated under conditions of cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
acute renal injury on the scale pRIFLE | 48 hours
  diagnosis of acute kidney injury after cardiac surgery

SECONDARY OUTCOMES:
TIMP-2 | 6 hours
  elevation of TIMP-2 after cardiac surgery
renal resistant index with doppler ultrasound | before, 6 hour, 24 hour
  with doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Siberian Biomedical Research Centre, Novosibirsk, Novosibirsk Oblast, Russia